CLINICAL TRIAL: NCT04582630
Title: Effects of Omega-3 Fatty Acids on Sarcopenia in Trauma Patients in Intensive Care Unit
Brief Title: Effects of Omega-3 Fatty Acids on Muscle Wasting
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hulya ULUSOY, Clinical Professor, Karadeniz Technical University
Other Study IDs: Karadeniz TU
Record Dates: First submitted 2020-07-22; First posted 2020-10-09 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Muscle Wasting
Keywords: Critical Illness; Trauma; Fatty Acids; Anthropometry; Nutrition Disorders; Sarcopenia
MeSH Terms: conditions — Muscular Atrophy; Critical Illness; Wounds and Injuries; Nutrition Disorders; Sarcopenia | interventions — Fatty Acids, Omega-3; Eicosapentaenoic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — TNF-a, IL-6, TOS, P3NP levels in muscle wasting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Omega 3 fatty acid: Participants will take 0.1-0.2 g/kg/day of omega 3 fatty acids for 7 days.
  Interventions: Dietary Supplement: omega 3 fatty acid
- Control (standart): Standart medical nutrition therapy

INTERVENTIONS:
Dietary Supplement: omega 3 fatty acid — Participants will take 0.1-0.2 g/kg/day of omega 3 fatty acids for 7 days.
  Other Names: eicosapentaenoic acid (EPA) and docosohexaenoic acid (DHA)
  Groups: Omega 3 fatty acid

SUMMARY:
The risk of muscle wasting, and sarcopenia is high in the intensive care unit patients and associated with adverse clinical outcomes. The etiology of muscle wasting is multifactorial and medical nutrition therapy plays a key role in treatment and prevention. The purpose of this study is to evaluate the effect of omega-3 fatty acids in the treatment and/or prevention of muscle wasting in critically ill trauma patients.

DETAILED DESCRIPTION:
Low skeletal muscle mass and loss of lean tissue in critically illness have been associated with negative clinical outcomes. Critically ill patients may lose about 25% of their skeletal muscle mass within 7 days of admission to the intensive care unit. Besides increased protein catabolism, other factors inherent to the ICU environment contribute to muscle loss, including patient immobility and interruptions in nutrient delivery. This combination of factors is especially debilitating in patients with preexisting low muscle stores due to sarcopenia, chronic illness, or malnutrition. Although preservation of skeletal muscle mass is important for recovery in critically ill patients, the mechanism of muscle wasting is not unknown. Muscle wasting is a multifactorial process and it may be the consequence of several events, including oxidative stress, inflammatory conditions and muscle remodeling. Omega-3 fatty acids with their anti-inflammatory, antioxidant and anabolic effects can be a key factor for an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years and ≤80 years, Expected ICU stay of seven days or longer Written informed consent or requirements of local/national ethical committee

Exclusion Criteria:

Pregnancy or breastfeeding Neuromuscular conditions (e.g., multiple sclerosis, muscular dystrophy, spinal cord injury, Guillain-Barre syndrome) Current cancer or chemotherapy End-stage of renal failure or dialysis treatment or renal transplantation prior to ICU admission Burn injury History of transplantation Pretibial edema Uncontrolled hemorrhage Uncontrolled hyperlipidemia Acute pancreatitis Acute thromboembolic diseases Severe heart failure Septic shock Concurrent enrolment in a nutrition-related interventional study at the time of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill trauma patients aged between 18 - 80 years of both sexes
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in rectus femoris muscle cross-sectional area | Baseline and 7 days
  Will be evaluated by ultrasound.
Changes in mid-upper arm and calf circumferences | Baseline and 7 days
  Will be measured by tape measure.
Changes in triceps and biceps skinfold thickness Changes in triceps and biceps skinfold thickness | Baseline and 7 days
  Will be measured by caliper.
Changes in biochemical parameters related to muscle homeostasis, oxidative stress and inflammation | Baseline and 7 days
  Biochemical parameters related to muscle wasting such as TNF-a, IL-6, TOS, P3NP

SECONDARY OUTCOMES:
Intensive care unit length of stay | Time of admission to the ICU until the time of discharge from the intensive care unit, up to 1 year
  Time from study inclusion to intensive care unit discharge.
Hospital Length of Stay | Time of discharge from the ICU until hospital discharge, up to 1 year
  Time from study inclusion to hospital discharge.
28-day mortality | 28 day
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Oguzhan Kucuk, MD, Principal Investigator — Karadeniz Technical University; Melda Kangalgil, MSc, Principal Investigator — Karadeniz Technical University; Kıvanc Oncu, MD, Principal Investigator — Karadeniz Technical University; Serap Ozer Yaman, PhD, Principal Investigator — Karadeniz Technical University; Sekine Turan, MD, Principal Investigator — Karadeniz Technical University; Süleyman Caner Karahan, MD, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University Medical Faculty Department of Anesthesiology and Reanimation, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No